CLINICAL TRIAL: NCT03849391
Title: Effect of Skate Skin Extract on Cognitive Function in Adults With Subjective Memory Impairment
Brief Title: Effect of Skate Skin Extract on Cognitive Function in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-2018-034
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Subjective Memory Impairment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skate group (Experimental): This group takes Skate Skin extract for 12 weeks
  Interventions: Dietary Supplement: Skate group
- Placebo group (Placebo Comparator): This group takes Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Skate group — This group takes 500 mg/day Skate Skin extract for 12 weeks
  Arms: Skate group
Dietary Supplement: Placebo group — This group takes 500 mg/day Placebo for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Skate Skin extract on cognitive function in adults with subjective memory impairment for 12 weeks.

DETAILED DESCRIPTION:
Previous animal studies have indicated that Skate Skin extract may have the ability to improve cognitive function. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Skate Skin extract on cognitive function in adults with subjective memory impairment for 12 weeks; the safety of the compound are also evaluate. The Investigators examine chemical and metabolic parameters, and cognitive function at baseline, as well as after 6 and 12 weeks of intervention. One hundred adults were administered either 500 mg of Skate Skin extract or a placebo each day for 12 weeks;

ELIGIBILITY:
Inclusion Criteria:

* Global Deterioration Scale (GDS) 2 or 3

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 3 times of upper limit of reference range and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of viral hepatitis or cancer
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination total score | Change from Baseline Mini-Mental State Examination total score at 3 months
  Change in Mini-Mental State Examination total score during 3 months

SECONDARY OUTCOMES:
Korean instrumental activity of daily living total score | Change from Baseline Korean instrumental activity of daily living total score at 3 months
  Change in Korean instrumental activity of daily living total score during 3 months
Computerized NeuroCognitive Function test total score | Change from Baseline Computerized NeuroCognitive Function test total score at 3 months
  Change in Computerized NeuroCognitive Function test total score during 3 months
brain derived neurotrophic factor | Change from Baseline brain derived neurotrophic factor level at 3 months
  Change in brain derived neurotrophic factor level during 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Integrated Research Institute for Natural Ingredients and Functional Foods, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided